CLINICAL TRIAL: NCT04120493
Title: A Phase 1/2, Randomized, Double-Blind, Sham Control and Open-Label Study to Explore Safety, Tolerability, and Efficacy Signals of Multiple Doses of Striatally-Administered rAAV5-miHTT Total Huntingtin Gene (HTT) Lowering Therapy (AMT-130) in Early Manifest Huntington's Disease
Brief Title: Safety and Proof-of-Concept (POC) Study With AMT-130 in Adults With Early Manifest Huntington's Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UniQure Biopharma B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-AMT-130-01
Record Dates: First submitted 2019-09-30; First posted 2019-10-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Huntington's Disease
Keywords: Gene therapy; AAV (adeno-associated virus); serotype 5 AAV (adeno-associated virus); serotype 5; Viral vector; miHTT; muHTT; Huntington's Disease (HD)
MeSH Terms: conditions — Huntington Disease | interventions — salicylhydroxamic acid; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Low dose rAAV5-miHTT (6x10^12 gc/subject).
  Note: gc = genome copies
  Interventions: Genetic: intra-striatal rAAV5-miHTT
- Cohort 2 (Experimental): High dose rAAV5-miHTT (6x10^13 gc/subject).
  Interventions: Genetic: intra-striatal rAAV5-miHTT
- Cohorts 1, 2 (Sham Comparator): Imitation (sham) surgery
  Interventions: Other: Imitation (sham) surgery
- Cohort 3 (Experimental): Low dose rAAV5-miHTT (6x10^12 gc/subject).
  High dose rAAV5-miHTT (6x10^13 gc/subject).
  Interventions: Genetic: intra-striatal rAAV5-miHTT
- Cohort 4 (Experimental): High dose rAAV5-miHTT (6x10^13 gc/subject).
  Interventions: Genetic: intra-striatal rAAV5-miHTT

INTERVENTIONS:
Genetic: intra-striatal rAAV5-miHTT — One time MRI-guided stereotaxic infusion of rAAV5-miHTT into the brain
  Other Names: AMT-130
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Other: Imitation (sham) surgery — Simulated surgical procedure with skin incisions only; no intrastriatal injections and no burr holes through the skull
  Arms: Cohorts 1, 2

SUMMARY:
This is the first study of AMT-130 in patients with early manifest HD and is designed to establish safety and proof-of-concept (PoC). CT-AMT-130-01 is a Phase 1/2, multicenter, first-in-human (FIH) study. The first three cohorts of the study have completed enrollment, including the randomized, double-blind, sham-controlled cohorts. Cohort 4 is open-label.

Cohort 4 participants will receive high dose AMT-130.

DETAILED DESCRIPTION:
AMT-130 is an investigational, single administration gene therapy intended to modify the disease course for HD. Preclinical studies have shown that AMT-130 lowers huntingtin protein and is associated with decreased progression of Huntington's Disease signs in animal models.

Cohort 1, 2, and 3 evaluated low dose and high dose AMT-130.

Cohort 4 will further evaluate the safety of high dose AMT-130 in participants with low striatal volume. All participants in Cohort 4 will receive high dose AMT-130 and will receive pre- and post-operative dexamethasone.

Cohorts 1 and 2 participants continue follow-up visits through 6 years after receipt of AMT-130. Cohorts 3 and 4 participants continue follow-up visits through 5 years after receipt of AMT-130.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent prior to the study and study-related procedure
* Participants 25 to 65 years of age of both sexes
* Cohorts 1, 2, & 4: Early manifest HD as defined by a UHDRS total functional capacity (TFC) score of 9 to 13 and EITHER a diagnostic confidence level (DCL) of 4 OR a DCL of 3 if the subject either meets the definition of multidimensional manifest HD (UHDRS question 80) or has cognitive symptoms
* Cohort 3: Early manifest HD as defined by a UHDRS TFC score of ≥ 11 and EITHER a DCL of 4 or a DCL of 3 with either a positive "Yes" response to UHDRS Question 80 (multidimensional manifest diagnosis on motor, cognitive, behavioral, functional) or DSM5 criteria for cognitive disorder (Movement Disorder Society Task Force criteria).
* HTT gene expansion testing with the presence of ≥40 CAG repeats
* Striatal MRI volume requirements per hemisphere:
* Cohorts 1, 2, & 3: Putamen ≥2.5 cm^3 (per side); Caudate ≥2.0 cm^3 (per side)
* Cohort 4: Putamen <2.5 cm^3 (on either side); Caudate <2.0 cm^3 (on either side)
* All HD concomitant medications (addressing motor, behavioral, and cognitive symptoms) must be stable for 3 months prior to Screening with no change in clinical symptoms requiring change in medication prior to anticipated administration procedure
* Able and willing to comply with all procedures and the study visit schedule as outlined in the protocol
* All female participants of childbearing potential (FOCP) must have a negative serum pregnancy test at Screening, (and Visit 1A, as appropriate), a negative pregnancy urine dipstick at Baseline, and not be breastfeeding. All FOCPs and sexually mature males must be compliant with a highly effective birth control method.

Exclusion Criteria:

* Evidence of suicide risk
* Receipt of an experimental agent within 60 days or five half-lives prior to Screening or anytime over the duration of this study.
* Participation in an investigational trial or investigational paradigm (such as exercise/physical activity, cognitive therapy, brain stimulation) within 60 days prior to Screening or anytime over the duration of this study.
* Presence of an implanted deep brain stimulation device, ventriculoperitoneal or other CSF shunt, or other implanted catheter
* Any history of gene therapy, RNA or DNA targeted HD specific investigational agents, such as antisense oligonucleotides (ASOs), cell transplantation or any other experimental brain surgery.
* Any contraindication to 3.0 Tesla MRI as per local guidelines
* Brain and spinal pathology that may interfere with the surgical delivery of AMT-130 or represents a significant neurologic comorbid disorder
* Any contraindication to lumbar puncture as per local guidelines
* Malignancy within 5 years of Screening, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
* Hospitalization for any major medical or surgical procedure involving general anesthesia within 12 weeks of Screening or planned during the study
* Current or recurrent disease, (including pre-existing cardiovascular or pulmonary conditions) infection, or other significant concurrent medical condition or medications that could confound clinical and laboratory evaluations or could affect a participant's safety or their ability to undergo the neurosurgical procedure or comply with the procedures and study visit schedule
* Known or suspected intolerance or hypersensitivity to the investigational product(s), closely-related compounds, or any of the stated ingredients
* Any known allergy to gadoteridol (ProHance)
* Screening laboratory values (as measured by the central laboratory): a. Alanine aminotransferase (ALT) >2 × upper limit of normal (ULN) b. Aspartate aminotransferase (AST) >2 × ULN c. Total bilirubin >2 × ULN d. Alkaline phosphatase (ALP) >2 × ULN e. Creatinine >1.5 × ULN f. Platelet count <100,000/mm3g.Prothrombin time (PT) >1.2 × ULN h. Partial thromboplastin time (PTT) >1.2 × ULN
* Known allergy, sensitivity, or other contraindication to medications in the immunosuppression regimen in this protocol.
* Any participant with an active infection (e.g., coronavirus disease 2019 [COVID-19]) at Screening or at the time of treatment that requires medical intervention. Participants may rescreen, or if screened eligible and an open surgical slot is available, may receive treatment after recovery.
* Cohort 4 ONLY: Inability to establish a safe trajectory to administer AMT-130 to the target structures, as assessed by neuroimaging.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number and type of Adverse Events (AE) | 12 months (Cohorts 1 & 2) and 12 months (Cohort 3)
  Safety will be assessed by adverse events (AEs) related to clinical safety laboratory tests, vital signs, electrocardiograms (ECGs), neurological and physical examinations, rAAV5 vector shedding, immunogenicity response (Cohorts 1, 2 & 3), suicidality risk [Columbia-Suicide Severity Rating Scale [C-SSRS)], changes in global cognitive functioning [Montreal Cognitive Assessment Scale (MoCA)] and MRI measures of edema, inflammation, volume loss and structural changes.

SECONDARY OUTCOMES:
Duration of persistence of AMT-130 in the brain | Collected for duration of study through month 72 (Cohorts 1 & 2) and through month 16 (Cohorts 3 & 4)
  Change over time in levels of AMT-130-derived Vector DNA Expression in the Cerebrospinal Fluid (CSF)

OTHER OUTCOMES:
CSF Mutant Protein (fM) | Collected for duration of study through month 72
  Will be used as an exploratory biomarker to measure disease progression and responsiveness to AMT-130 treatment.
CSF/Serum Neurofilament Light Chain (pg/mL) | Collected for duration of study through month 72
  Will be used as an exploratory biomarker to measure disease progression and responsiveness to AMT-130 treatment.
Unified Huntington Disease Rating Scale (UHDRS) | Collected for duration of study through month 72
  The UHDRS will assess changes from baseline in summary scores of domains of motor function, cognitive function, behavioral function, and functional abilities.
Quantitative Motor (Q-Motor) Testing | Collected for duration of study through month 72 (Cohorts 1, 2 & 3)
  Q-Motor testing will measure disease progression and responsiveness to AMT-130 treatment.
Magnetic Resonance Imaging (MRI) | Collected for duration of study through month 72
  MRI assessments will include whole brain volume, striatal region volumes, white matter volume, gray matter volume, ventricular volume, cortical thickness, and diffusion MRI measures.
Neuro-QoL Measures | Collected for duration of study through month 72
  The Neuro-QoL is a brief, reliable, valid, standardized set of patient reported, Health Related Quality of Life (HRQoL) measures for people living with neurological conditions.

CONTACTS AND LOCATIONS:
Overall Officials: David H. Margolin, MD, PhD, Study Director — uniQure, Inc.
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona (Surgical Site Only), Tucson, Arizona
  - University of California, San Francisco, San Francisco, California
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Department of Neurology, Ann Arbor, Michigan
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas, Houston, Texas
  - Virginia Commonwealth University VCU School of Medicine, Department of Neurology, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pala M, Yilmaz SG. Circular RNAs, miRNAs, and Exosomes: Their Roles and Importance in Amyloid-Beta and Tau Pathologies in Alzheimer's Disease. Neural Plast. 2025 Apr 8;2025:9581369. doi: 10.1155/np/9581369. eCollection 2025. PMID 40235521
- [Derived] Estevez-Fraga C, Tabrizi SJ, Wild EJ. Huntington's Disease Clinical Trials Corner: March 2024. J Huntingtons Dis. 2024;13(1):1-14. doi: 10.3233/JHD-240017. PMID 38489195
- [Derived] Estevez-Fraga C, Tabrizi SJ, Wild EJ. Huntington's Disease Clinical Trials Corner: November 2022. J Huntingtons Dis. 2022;11(4):351-367. doi: 10.3233/JHD-229006. PMID 36463457
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: April 2020. J Huntingtons Dis. 2020;9(2):185-197. doi: 10.3233/JHD-200002. PMID 32250312